CLINICAL TRIAL: NCT01189903
Title: Clinical Evaluation - A Phase IIA Proof of Concept Study of Regorafenib (Bayer 73-4506) in Biopsy-amenable Asian Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Purpose: Treatment
Other Study IDs: CR01/18/10
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Asian Colorectal Cancer Patients
MeSH Terms: interventions — regorafenib

INTERVENTIONS:
Drug: Regorafenib

SUMMARY:
1. Primary Endpoints

   * Biomarker data suggestive of regorafenib-mediated inhibition of the RAS-RAF- MEK-ERK signal transduction pathway,of various tyrosine kinase receptors and/or of angiogenesis.
   * Evaluation of potential relationships between biomarker data and clinical activity.
   * Evaluation of a novel biomarker technology (Prometheus COPIA platform)
2. Secondary Endpoints

   * Biomarker data suggestive of regorafenib-mediated effects on circulating rare cells.
   * Comparison of tumor genetic profiles obtained using DNA isolated from plasma, tumor biopsies and circulating tumor cells.
   * Patient safety data
   * Pharmacokinetics of regorafenib
   * Changes in tumor metabolic activity as measured by PET CT scan (optional)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven metastatic colorectal adenocarcinoma that is refractory to standard therapy and not amenable to surgery with curative intent.
* Tumor characteristics:

  * At least one lesion that is suitable for a repeated biopsy; eg. subcutaneous nodule, skin lesion, rectal tumor, colonic mass easily reached by colonoscopy, peritoneal masses at least 3cm in maximum diameter that are easily assessable by image guided core biopsy.
  * For liver lesions, more superficially located lesions at least 3cm in maximum dimension with a rim of normal liver tissue, assessable safely by image guided core biopsy as determined by an experienced interventional radiologist.
* Eastern Cooperative Oncology Group ECOG performance status of 0 or 1 (see Appendix 10.4).
* Adequate bone marrow function (absolute neutrophil count =1,500/mm3; platelet count =100000/mm3; hemoglobin =9g/dl
* Adequate liver and renal function as assessed by the following laboratory requirements conducted within 7 days of starting to study treatment:

  * Total bilirubin < 1.5 x the upper limit of normal (ULN).
  * Alanine transaminase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN (< 5 x ULN for patients with liver involvement of their cancer).
  * Amylase and lipase < 1.5 x the ULN
  * Serum creatinine < 1.5 x the ULN.
  * Glomerular filtration rate (GFR) = 30 ml/min/1.73 m2 according to the MDRD (Modified diet in renal disease) abbreviated formula
* Prothrombin time, international normalized ratio (INR) and partial thromboplastin time less than or equal to 1.2 times the ULN.
* Male or female at least 21 years of age.
* A female subject is eligible to enter and participate in the study if she is:

  * Non-childbearing potential (ie. physiologically incapable of becoming pregnant) including any women who:
  * Has had a hysterectomy or
  * Has bilateral oophorectomy (ovariectomy) or
  * Has bilateral tubal ligation or
  * Is postmenopausal (demonstrate total cessation of menses for greater than or
  * Childbearing potential, has a negative serum or urine pregnancy test at screening, agrees to one of the following: double barrier contraception or abstinence.
* Predicted life expectancy of at least 12 weeks.
* Resting oxygen saturation greater than 92% on room air.
* Written informed consent.
* Able to swallow and retain oral medication.
* Prothrombin time (PT), International Normalized Ratio for PT (PT INR), and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) within normal limits.

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-01; Primary Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Goh BC, Fleming GF, Janisch L, Vogelzang NJ, Stadler WM, Ratain MJ. Development of a schedule-dependent population pharmacodynamic model for rhizoxin without quantitation of plasma concentrations. Cancer Chemother Pharmacol. 2000;45(6):489-94. doi: 10.1007/s002800051024. PMID 10854137
- [Background] Vokes EE, Goh BC, Bertucci D, Vogelzang NJ, Mani S, Ratain MJ. A Phase I study of raltitrexed and paclitaxel given every 3 weeks to patients with solid tumors. Cancer. 1999 Aug 1;86(3):528-32. PMID 10430263